CLINICAL TRIAL: NCT06915779
Title: Long Term Follow-up Study of CTN 236 - A Study of an HPV VLP Vaccine in a Cohort of HIV Positive Girls and Women
Brief Title: Long Term Follow-up of HPV Vaccine in HIV (CTN 236)
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network); Women's Health Research Institute of British Columbia (Other); Canadian Institutes of Health Research (CIHR) (Other Government); BC Women's Hospital & Health Centre (Other); Merck Canada Inc. (Industry); University Health Network, Toronto (Other); McGill University (Other); University of Saskatoon (Unknown); British Columbia Centre for Disease Control (Other Government); Vaccine Evaluation Center, Canada (Other); British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Deborah Money, Executive Vice Dean, Faculty of Medicine, Professor, Dept. OB/GYN, University of British Columbia
Other Study IDs: H14-02364
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Cervical Cancer; Human Papillomavirus Infection; Human Immunodeficiency Virus; Cervical Dysplasia; Genital Warts
Keywords: HPV; HPV Vaccine; HIV; Women; Genital Warts; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Acquired Immunodeficiency Syndrome; Uterine Cervical Dysplasia; Condylomata Acuminata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Cervical cytology and HPV DNA (liquid prep method) Gynecological swab for vaginal microbiota Serology for HPV antibodies Serology for HSV-2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: HIV positive girls and women (greater than, or equal to, age 11) attending the HIV treatment clinics in each of the 13 sites across Canada and who have enrolled in the original study, "A Study of an HPV VLP Vaccine in a Cohort of HIV Positive Girls and Women (CTN 236)" and received at least one dose of quadrivalent HPV vaccine, will be offered participation on this study.

SUMMARY:
The purpose of this extension study is to determine whether HPV antibody levels in HIV-positive girls and women will decline more rapidly and more significantly than in HIV-negative girls and women and if this decline is determined by HIV parameters.

DETAILED DESCRIPTION:
Study hypothesis: HPV antibody levels in HIV-positive girls and women will decline more rapidly and more significantly than in HIV-negative girls and women and that this decline will be determined by HIV parameters.

Girls and women living with HIV (greater than, or equal to, age 11) attending the HIV treatment clinics in each of the 13 sites across Canada and who enrolled in and received at least one dose of quadrivalent HPV vaccine as part of "A Study of an HPV VLP Vaccine in a Cohort of HIV Positive Girls and Women (CTN 236)" will be offered participation in this long term follow-up study.

OBJECTIVES

Primary:

To measure the antibody response to each genotype contained in the qHPV vaccine to 96 months post first dose of quadrivalent HPV vaccine.

Secondary:

1. To determine the incidence rate and nature of 'breakthrough' HPV incidence and persistent (2 sequential positive HPV DNA in > 6 months) infections of vaccine - non-vaccine-containing high-risk types;
2. To determine the incidence rate of cervical dysplasia (LSIL or greater) and/or vulvar and vaginal dysplasia associated HPV genotypes (both with and without vaccine types; and
3. To determine the incidence rate of external genital warts.

Exploratory:

1. To examine the relationship between HSV-2 serostatus and peak HPV antibody response as well as HPV incidence and persistent infections; and
2. To relate vaginal microbiome profiles to HPV acquisition/persistence and cervical dysplasia.

STUDY DESIGN Phase 3, longitudinal, multi-center, 13 sites, girls and women living with HIV aged 11 years of age and older, received one plus dose of quadrivalent HPV vaccine in the precursor study.

STUDY VISITS 3 possible visits over a total of 5 years

* Visit 8 (month 36)
* Visit 9 (month 48)
* Visit 10 (month 60)
* Visit 11 (month 72)*
* Visit 12 (month 84)*
* Visit 13 (month 96)*

STUDY PROCEDURES:

Informed consent, Medical history, Height & weight, Cervical cytology and HPV DNA (liquid prep method), Gynecological swab for vaginal microbiota, Serology for HPV antibodies, Serology for HSV-2, Lower Urinary Tract Symptoms Survey (at one time-point only for participants 18 years of age and older).

NOTE: Girls who are pre-menarchal and not sexually active will not be asked to undergo any genital examinations or sampling until they become menarchal and sexually active.

DATA COLLECTION Consent and source document templates will be provided by the Study Coordinating Center. Source data will be transferred to paper case report forms and sent to the Study Coordinating Center/CTN where it will be entered into an electronic database.

PRIMARY ENDPOINT The primary endpoint of this study will be the HPV antibody GMT for each of the 4 types contained in the GARDASIL™ vaccine up to month 96 after receiving at least one dose of the vaccine.

SECONDARY ENDPOINTS Incidence rates of: 1) breakthrough incidents and persistent HPV infections; 2) cervical dysplasia; 3) external genital warts

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in CTN 236 study, phase 1
* Able to give fully informed consent or assent

Exclusion Criteria:

* Did not receive at least one vaccination via CTN 236, phase 1
* Cannot provide fully informed consent or assent

Ages: 11 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV positive girls and women (greater than, or equal to, age 11) attending the HIV treatment clinics in each of the 13 sites across Canada and who have enrolled in the original study, "A Study of an HPV VLP Vaccine in a Cohort of HIV Positive Girls and Women (CTN 236)" and received at least one dose of the quadrivalent HPV vaccine, will be offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Primary Objective | 96 month post-vaccination regimen
  To measure the antibody response to each genotype contained in the qHPV vaccine to 96 months post-vaccination regimen.

SECONDARY OUTCOMES:
Secondary Objective #1 | 96 month post-vaccination regimen
  To determine the incidence rate and nature of 'breakthrough' HPV incidence and persistent (2 sequential positive HPV DNA in > 6 months) infections of vaccine - non-vaccine-containing high-risk types.
Secondary Objective #2 | 96 month post-vaccination regimen
  To determine the incidence rate of cervical dysplasia (LSIL or greater) and/or vulvar and vaginal dysplasia associated HPV genotypes (both with and without vaccine types
Secondary Objective #3 | 96 month post-vaccination regimen
  To determine the incidence rate of external genital warts.

OTHER OUTCOMES:
Exploratory Objective #1 | 96 month post-vaccination regimen
  To examine the relationship between HSV-2 serostatus and peak HPV antibody response as well as HPV incidence and persistent infections
Exploratory Objective #2 | 96 month post-vaccination regimen
  To relate vaginal microbiome profiles to HPV acquisition/persistence and cervical dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah M Money, MD, FRCSC, Principal Investigator — Dept. OB/GYN, University of British Columbia
Locations (13):
- Canada (13):
  - Oak Tree Clinic, BC Women's Hospital & Health Centre, Vancouver, British Columbia
  - AIDS Research Program & the John Ruedy Immunodeficience Clinic, St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - Infection & Immunology Clinic, Hotel Dieu, Kingston, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Maple Leaf Research, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - HIV Care Program, Windsor, Ontario
  - Centre de maternal et infantile sur le sida, CHU Sainte Justine, Montreal, Quebec
  - Chronic Viral Illness Service, Hopital Royal Victoria (McGill University), Montreal, Quebec
  - CHUL and Mother-Child Center Soleil, Centre de Recherche en Infectiologie CHU de Quebec, (Universite Laval), Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT06915779/Prot_SAP_000.pdf